CLINICAL TRIAL: NCT02253433
Title: The Houston Home-Based Integrated Intervention Targeting Better Asthma Control (HIITBAC) for African Americans
Brief Title: The Houston HIITBAC for African Americans
Acronym: HIIT-BAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Harris County Hospital District (Other Government); Houston Department of Health and Human Services (Unknown); Texas A&M University (Other); M.D. Anderson Cancer Center (Other); UTHealth School of Public Health (Unknown)
Responsible Party: Principal Investigator, Winifred J. Hamilton, PhD, Director, Environmental Health Service, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCORI AS-1308-05887; H-34115 (Other: Baylor College of Medicine)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Asthma
Keywords: asthma; environmental triggers; home-based intervention; asthma home visits
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Clinic Care (Experimental): This arm receives enhanced in-clinic care only.
  Interventions: Other: Enhanced Clinic Care
- Enhanced Clinic Care + Home Intervention (Experimental): This arm receives the enhanced in-clinic care intervention, as well as a home-based intervention.
  Interventions: Other: Enhanced Clinic Care; Other: Enhanced Clinic Care + Home Intervention

INTERVENTIONS:
Other: Enhanced Clinic Care — The intervention includes a standard clinical appointment including spirometry, as well as collection of self-report information from detailed health and exposure questionnaires, asthma education, assessment for allergies, and a customized asthma self-management plan developed using motivational interviewing.
Other: Enhanced Clinic Care + Home Intervention — The home-based component includes environmental exposure assessment (observed and measured) and a multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).
  Arms: Enhanced Clinic Care + Home Intervention

SUMMARY:
The purpose of this study is to improve the health of African-American adults who have poorly controlled asthma. The study compares a home-based exposure reduction and asthma control intervention to enhanced in-clinic care that includes a standard clinical appointment as well as information from a detailed exposure history, asthma education, assessment for allergies, and a customized asthma self-management plan developed using motivational interviewing. The interventional group receives enhanced in-clinic care, as well as a customized home-based environmental exposure assessment and multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).

DETAILED DESCRIPTION:
The study hypothesis is that the addition of a holistic, home-based environmental exposure reduction and asthma control intervention to enhanced in-clinic care will result in statistically significant improvements in key measures of health and quality of life among Houston-area African-American adults with poorly controlled asthma.

This is a pragmatic randomized controlled clinical trial that compares the effectiveness of a customized, holistic, patient-centered, home-based environmental intervention for improving asthma control (the "intervention") with enhanced clinic-based care. Both arms receive identical in-clinic care, including collected self-report information from detailed health and exposure questionnaires, asthma education, assessment for allergies, and a customized asthma self-management plan developed using motivational interviewing. The intent of the study is to assess-real-life effectiveness of a home-based intervention in African-American adults with poorly controlled asthma.

ELIGIBILITY:
INCLUSION CRITERIA:

* African-American
* 18 years of age or older
* Diagnosis of poorly controlled asthma*
* Fixed address within Harris County, Texas, with no intention of moving within the following 12 months
* Working telephone number
* Verbally fluent in English

  * Poorly controlled asthma was defined as (1) diagnosed by a physician as having asthma in the past and currently has asthma, and (2) fulfills one or more of the following criteria: (a) one or more emergency department (ED), urgent care visits or hospitalizations for asthma in the preceding year; (b) meets the definition of "very poorly controlled" asthma as defined by the National Asthma Education and Prevention Program, Third Expert Panel on the Diagnosis and Management of Asthma (definition includes daily asthma symptoms, nighttime awakenings two or more times per week, extremely limited normal activity, and/or daily use of a short-acting beta agonist for symptom control); and/or (c) an Asthma Control Test score of 19 or lower.

EXCLUSION CRITERIA:

* Severe co-morbid conditions-such as a poorly controlled psychiatric illness or a condition requiring intense medical treatment that could reasonably be expected to (1) confound the effects of this study's intervention, (2) make it unlikely that a participant could follow the treatment plan, or (3) pose a safety issue for the home-visit team.
* A concurrent pulmonary study that could reasonably be expected to confound the effects of the intervention.
* Living in a group living facility, such as a nursing home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winifred J Hamilton, PhD, SM, Principal Investigator — Baylor College of Medicine
Locations (1):
- Harris Health Smith Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants receive their individual laboratory, exposure and other data, as well as their customized asthma control plan, to help them manage their asthma. This information is delivered to participants at clinic and/or at home visits as appropriate. Laboratory results may be mailed as well. Aggregate data were made available to participants at a regional Town Hall 5/1/2018 and by mail as requested at exit by participants. Aggregate and/or de-identified data were and are being made available to the Patient / Stakeholder Advisory Board and to researchers through presentations, websites, publications and data sharing arrangements. No identifiable IDP will be made available to other researchers except through consent of the participant and IRB approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The study protocol and ICF have been shared and are available on request. At the aggregate level, the initial findings of the pragmatic clinical trial were made available to our Patient/Stakeholder Advisory Panel at the February 12, 2018 meeting of the panel; at a regional Town Hall on asthma on May 1, 2018; and to participants who requested results by mail in November 2018. The Draft Final Research Report was submitted to PCORI in September 2018 and is undergoing external peer review. Two manuscripts--on methods and initial results--are being finalized for journal submission. The SAP and analytic code are currently undergoing refinement as we begin our secondary analyses and should be available in 2019.
Access Criteria: Access criteria are based on protection of individual participant data as described in the protocol and ICF. Aggregate and de-identified data will be made available electronically, in the Rice University Kinder Urban Data Base Platform, and in presentations and manuscripts.
URL: https://www.bcm.edu/environmentalhealth

REFERENCES:
- [Derived] Bruhl RJ, Perkison WB, Hanania NA, McNeill LH, Oluyomi AO, Fiesinger EB, Minard CG, Solomon A, Hamilton WJ; Patient/Stakeholder Advisory Board and other members of the HIITBAC Research Team:; Butler B, Caldwell J, Crosby E, Davis C, Galvan H, Harris R, Lacour-Chestnut F, Martin C, Pannell S, Phipps K, Richardson G, Solomon A, White W, Boles J, Rangel A, Virk R, Brock M, Guffey D, Ramamurthy U, Persse D, Maffei S, Chan W, Reyes B. Design of a home-based intervention for Houston-area African-American adults with asthma: Methods and lessons learned from a pragmatic randomized trial. Contemp Clin Trials. 2020 Apr;91:105977. doi: 10.1016/j.cct.2020.105977. Epub 2020 Mar 6. PMID 32151753

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Clinic Care: This arm will receive enhanced in-clinic care that includes a standard clinical appointment as well as information from a detailed exposure history, asthma education, assessment for allergies, and a customized asthma self-management plan developed using motivational interviewing.
- Enhanced Clinic Care + Home Intervention: This arm receives enhanced in-clinic care, as well as a customized home-based environmental exposure assessment and multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).
  Enhanced in-clinic care and intervention: This arm receives enhanced in-clinic care, as well as a customized home-based environmental exposure assessment and multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).
Period: Overall Study
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Home Intervention
Started | 130 | 134
Completed | 114 | 79
Not Completed | 16 | 55
Not completed — Unable to Contact | 9 | 16
Not completed — Death | 1 | 1
Not completed — No Longer Interested | 3 | 15
Not completed — Out of Study Area | 2 | 7
Not completed — Uncomfortable with home visitors | 0 | 3
Not completed — Unstable Housing/Homeless | 0 | 7
Not completed — Too Busy | 0 | 4
Not completed — Medical or Other Concerns | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Home Intervention | Total
Number analyzed (Participants) | 130 | 134 | 264
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 117 | 118 | 235
  >=65 years | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.7) | 51.0 (13.3) | 50.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 98 | 196
  Male | 32 | 36 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 130 | 134 | 264
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 130 | 134 | 264
Asthma Control Test (ACT) [Mean (Standard Deviation); unit: units on a scale] — The ACT is a validated 5-question scale assessing asthma control over the previous four weeks. Each question has five possible responses, from 1 (worst) to 5 (best). The total score ranges from 5 (worst control) to 25 (best control). In general, a total score of 19 or less suggests poor control. Population: One participant consented and withdrew before any baseline characteristics (aside from age, gender and race) were collected. A second participant chose not to answer all five questions.
  units on a scale
    number analyzed (Participants) | 129 | 133 | 262
    (all) | 12.5 (4.3) | 12.5 (4.2) | 12.5 (4.3)
Juniper Mini Asthma Quality of Life Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Self report. A validated 15-item questionnaire, with each question having seven possible answers score from 1 (worst) to 7 (best). Minimum total score is 15 (worst asthma quality of life). Maximum total score is 105 (best asthma quality of life). By design, an individual's score is reported as the mean (total score/15). Thus the possible mean reported score ranges from 1 (worst asthma quality of life) to 7 (best asthma quality of life). Population: In the enhanced clinical care ("control") group, one person withdrew immediately after consent, and two individuals chose not to answer one of the 15 questions. In the home-visit ("intervention") group, three individuals chose not to answer one question. Interpolation (inserted worst answer) was used in some of the analyses.
  units on a scale
    number analyzed (Participants) | 127 | 131 | 258
    (all) | 3.3 (1.2) | 3.2 (1.1) | 3.2 (1.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Measured at clinic. BMI = weight (kilograms) divided by height (meters) squared. It is an estimate of body fat in adults. 30 and higher = obese. Population: One person withdrew immediately after consent.
  kg/m^2
    number analyzed (Participants) | 129 | 134 | 263
    (all) | 36.0 (10.6) | 34.4 (10.1) | 35.2 (10.4)
Total Immunoglobulin E (Total IgE) [Mean (Standard Deviation); unit: kU/L] — Total IgE is a measure of the immunoglobulin E antibody in the blood, and an estimate of allergic status. The laboratory lowest level of detection was 18 kU/L. Guidelines vary and must be assessed in conjunction with clinical presentation and allergen-specific testing, but for this population we consider a Total IgE > 100 kU/L to be of clinical relevance. Population: One participant withdrew immediately after consent, permission for a blood draw was not given by two patients, and blood could not be obtained or was insufficient for analysis in four patients.
  kU/L
    number analyzed (Participants) | 127 | 131 | 258
    (all) | 550.5 (1479.8) | 643.2 (1217.6) | 597.6 (1351.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control Test (ACT) Score
Description: Self report. The ACT is a validated 5-question scale assessing asthma control over the previous four weeks. Each question has five possible responses, from 1 (worst) to 5 (best). The total score ranges from 5 (worst control) to 25 (best control). In general, a total score of 19 or less suggests poor control.
Time Frame: At baseline (enrollment) and exit (approximately 12 mo after enrollment)
Population: At baseline, one individual in each group chose not to answer all five ACT questions; therefore a total ACT score could not be calculated for those two individuals (missing data are addressed in the analyses). At exit, among those who completed the study, one person in the enhanced in-clinic group chose not to answer all five ACT questions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Home Intervention
Number analyzed (Participants) | 130 | 134
score on a scale
  Baseline: number analyzed (Participants) | 129 | 133
  Baseline | 12.5 (4.3) | 12.5 (4.2)
  Exit: number analyzed (Participants) | 113 | 79
  Exit | 16.2 (5.1) | 16.8 (5.1)
Statistical Analysis 1: Comparison: Enhanced Clinic Care vs Enhanced Clinic Care + Home Intervention; Test type: Superiority; p = 0.575, Mixed Models Analysis; Mean Difference (Final Values) = .60, 95% CI 2-sided [-.87 to 2.07]

2. Primary Outcome: Change in Juniper Mini Asthma Quality of Life Questionnaire Score (MiniAQLQ)
Description: Self report. A validated 15-item questionnaire, with each question having seven possible answers score from 1 (worst) to 7 (best). Minimum total score is 15 (worst asthma quality of life). Maximum total score is 105 (best asthma quality of life). By design, an individual's score is reported as the mean (total score/15). Thus the possible mean reported score ranges from 1 (worst asthma quality of life) to 7 (best asthma quality of life).
Time Frame: At baseline (enrollment) and exit (approximately 12 mo after enrollment)
Population: Among the enhanced in-clinic care group, one person withdrew immediately after consent and two individuals chose not to fill out all of the answers, such that a score could not be computer. At exit, 3 control and 1 intervention were missing (1) or incomplete (3).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Home Intervention
Number analyzed (Participants) | 127 | 134
score on a scale
  Baseline | 3.3 (1.2) | 3.2 (1.1)
  Exit: number analyzed (Participants) | 111 | 77
  Exit | 4.3 (1.5) | 4.5 (1.5)
Statistical Analysis 1: Comparison: Enhanced Clinic Care vs Enhanced Clinic Care + Home Intervention; Test type: Superiority; p = 0.141, Mixed Models Analysis; Mean Difference (Final Values) = .25, 95% CI 2-sided [-.18 to .68]

3. Secondary Outcome: Change in Emergency Department (ED) Visits for Asthma
Description: Self report. The healthcare utilization questions were from the validated CDC-BRFSS Asthma Survey. For this outcome measure, we used patient responses to a question that asked "During the past 12 months, how many times to you visit an emergency room of urgent care center because of your asthma?". We collected this information for the 12 months preceding their baseline and exit clinic visits. A higher number of visits suggests poorer asthma control.
Time Frame: At baseline (enrollment) and exit (approximately 12 mo after enrollment)
Population: One patient from the enhanced in-clinic only group withdrew immediately after consenting.114 "control" and 79 "intervention" completed the study. Respondent number less than enrollment and/or exit numbers reflects individuals who chose not to respond to the question.
Measure: Mean (Standard Deviation); unit: visits
Groups:
- Enhanced Clinic Care + Intervention: This arm receives enhanced in-clinic care, as well as a customized home-based environmental exposure assessment and multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).
  Enhanced in-clinic care and intervention: This arm receives enhanced in-clinic care, as well as a customized home-based environmental exposure assessment and multicomponent exposure reduction and asthma control intervention (five home visits over approximately 12 months).
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Intervention
Number analyzed (Participants) | 130 | 134
visits
  Baseline: number analyzed (Participants) | 120 | 129
  Baseline | 2.2 (3.5) | 2.6 (3.5)
  Exit: number analyzed (Participants) | 109 | 78
  Exit | 1.3 (2.4) | 1.1 (2.0)
Statistical Analysis 1: Comparison: Enhanced Clinic Care vs Enhanced Clinic Care + Intervention; Test type: Superiority; p = 0.043, Mixed Models Analysis; ED visits over the previous 12 months were positively skewed (skewness 2.95; kurtosis 14.1); the responses were dichotomized (0 vs. 1 or more); Odds Ratio (OR) = .86, 95% CI 2-sided [.47 to 1.57]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Enhanced Clinic Care | Enhanced Clinic Care + Home Intervention
All-Cause Mortality (participants affected / at risk) | 1/130 | 1/134
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/134
Other Adverse Events (participants affected / at risk) | 0/130 | 0/134

LIMITATIONS AND CAVEATS:
Limitations included (1) lack of a control group (the enhanced clinic visit = a robust intervention), (2) mobility of the participants, (3) disproportionate lost to follow-up, (4) missing data, (5) out-of-window encounters, and (6) Hurricane Harvey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT02253433/Prot_000.pdf
  • Informed Consent Form (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT02253433/ICF_001.pdf
  • Statistical Analysis Plan (2018-09-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02253433/SAP_002.pdf